CLINICAL TRIAL: NCT04964011
Title: Board Game Intervention to Improve Cognitive and Daily Functioning in Elderly People With Mild Cognitive Impairment: A Randomized Controlled Trial
Brief Title: Board Game Intervention to Improve Cognitive and Daily Functioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yang Shang-Yu (Other)
Responsible Party: Sponsor-Investigator, Yang Shang-Yu, Assistant professor, National Cheng Kung University
Organization: National Cheng Kung University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: CRREC-108-141
Record Dates: First submitted 2021-07-04; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Board game group (Experimental): The Board game group was led by an occupational therapist who has been working for six years. The intervention comprised 1 week of board game instruction and 11 weeks of board game tasks (combined with daily tasks), for a total of 12 weeks, once a week for 2 hours, for a total of 24 hours of intervention.
  Interventions: Other: Board game intervention
- Health promotion group (Active Comparator): MCI seniors in the health promotion group received general health promotion and were led by instructors from the long-term care facility for 12 weeks, including 4 weeks of physical activities, 4 weeks of singing activities, and 4 weeks of art activities, once a week for 2 hours, for a total of 24 hours.
  Interventions: Other: Board game intervention

INTERVENTIONS:
Other: Board game intervention — In this study, the two groups, the Board game group (12-week board game intervention) and Health promotion group (12-week general health promotion intervention).

SUMMARY:
Background:

With the rapid rise of the aging population, the number of seniors with mild cognitive impairment (MCI) has increased, and without timely interventions, participants are at high risk of developing dementia. Board games have become a popular tool for cognitive training, but many board games may not be appropriate for seniors and lack the support of empirical research.

Objectives:

To examine the effectiveness of a 12-week board game intervention for MCI seniors in improving cognitive functioning and scores on the instrumental activities of daily living (IADL) scale.

Methods:

A single-blind randomized controlled trial was conducted to collect data from a long-term care facility in central Taiwan. Sixty-eight MCI seniors were recruited and randomized into a board game group (trial group) and a health promotion group (control group). Participants in both groups received a 2-hour intervention once a week for 12 weeks, with the trial group receiving 12 weeks of board games and the control group receiving 12 weeks of health promotion activities. Before and after the intervention, the primary assessment was conducted using the Saint Louis University Mental Status Exam, Contextual Memory Test, and Trail Making Test part-A; the secondary assessment was conducted using the IADL scale.

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years or older without a diagnosis of dementia
* mild neurocognitive impairment

Exclusion Criteria:

* non-national senior citizens
* unable to understand the content and complete the questionnaire
* unable to participate in the full 12-week intervention
* had an acute illness such as a cold during the trial.

Ages: 65 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-01-03 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Saint Louis University Mental Status Exam (SLUMSE) | 15-25 minutes
  SLUMSE was used to evaluate the cognitive function of MCI seniors. SLUMSE is the most popular cognitive screening tool used worldwide to detect patients with dementia and MCI. The scale is comprised of four domains: orientation (e.g., day, year, and place; three questions), memory (e.g., remembering five things; one question), attention (e.g., story review; one question), and executive function (e.g., number counting, animal naming, picture recognition, size discrimination, and clock drawing; five questions). It contains 11 assessment items, with a total score of 0-30. A higher score indicates a higher level of cognition (Tariq, Tumosa, Chibnall, Perry III, & Morley, 2006).
Contextual Memory Test (CMT) | 15-20 minutes
  The CMT Memory Subscale was used to assess the memory function of MCI seniors. The CMT, a standardized memory assessment tool developed by Toglia (1993) for occupational therapists, was used to assess individual memory and meta-memory functions. This test consists of 2 cards with 20 items each related to a restaurant or breakfast (Tsai, 2006). Each card is divided into 3 dimensions: the recall subscale (40 questions), the recall awareness subscale (7 questions), and the memory strategy use subscale (6 questions). Only the recall subscale was used in this study, which included 2 dimensions: immediate recall (20 questions) and delayed recall (20 questions). Immediate recall is the ability to recall information that was accessed within 60 seconds; delayed recall is the ability to recall information that was accessed several minutes or hours ago. The total score for both immediate recall and delayed recall was 0-20, with higher scores indicating better recall ability.
Trail Making Test part-A (TMT-A) | 15-20 minutes
  The TMT-A, designed by Partington (1949), was used to assess the focused attention, selective attention, and executive function of MCI seniors. The participants were recorded in terms of reaction time (in seconds), starting with the number 1 and continuing sequentially until the number 25. The test was scored based on the time required to complete the connection, with lower scores indicating better ability (Tombaugh, 2004). This test has good reliability and validity (Kuo, 2018).

SECONDARY OUTCOMES:
Instrumental activities of daily living (IADL) | 10-20 minutes
  The IADL was used to assess IADL function in MCI seniors. The IADL is an eight-question scale developed by Lawton, Brody, and Médecin (1969). This scale is used to assess the ability to maintain independence, which is more complex than the average individual's self-care needs. The IADL is divided into eight dimensions, including cooking, shopping, going out, housekeeping, doing laundry, making phone calls, taking medication, and managing finances. Those who check 1 or 0 are classified as disabled, with a total score of 0-8. In addition, those who need assistance with three or more of the five items (i.e., shopping, going out, cooking, housekeeping, and doing laundry) are considered mildly disabled with a score of 5 or less. The scale has good reliability and validity (Chang, Hsieh, Hsueh, & Hsieh, 2006).

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Univeraity, Taichung, WuFeng, Taiwan